CLINICAL TRIAL: NCT06722924
Title: Definition of Acute Kidney Injury Based on Urine Output
Brief Title: Definition of Acute Kidney Injury by Urine Output in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: AKI-UO
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; Critical Illness; Critical Care, Intensive Care; Critical Care, Fluid Resuscitation
Keywords: observational study
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the association between urine output and acute kidney injury in severely ill patients admitted to intensive care units. The main research questions are:

What is the optimal threshold for defining reduced urine output in critically ill patients in intensive care? Is this threshold the same for different outcomes such as acute kidney injury, chronic kidney dysfunction, or mortality? Does this threshold change with treatment involving diuretics or dialysis? Does the patient's fluid balance or the amount of administered fluid affect the association between reduced urine output and the outcomes mentioned above? Is the optimal threshold for defining reduced urine output different for various patient categories and diagnoses, such as sepsis, burn injuries, or ARDS? Are there differences between surgical and non-surgical patients regarding the optimal threshold for defining reduced urine output in intensive care? Does the patient's comorbidity influence the level of reduced urine output that should be considered pathological?

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a common occurrence in critically ill patients in intensive care units and is strongly associated with an increased risk of complications, longer hospital stay and mortality. Research in this area was long hampered by the lack of a unified definition, but since 2012, there has been a widely accepted consensus definition for AKI: the KDIGO Clinical Practice Guideline for Acute Kidney Injury. This has facilitated comparisons of different studies and interventions.

According to this definition, AKI is based on either a) an acute elevation in blood creatinine levels (a breakdown product normally excreted in the urine) and/or b) reduced urine output. Kidney injury is further graded into three stages (1-3) based on increasing creatinine levels or decreasing urine output, where higher stages indicate worse kidney function and an increased risk of mortality.

However, the current definition of AKI also has weaknesses and limitations. Creatinine, a breakdown product primarily produced in the muscles, increases in the blood with kidney injury but reflects not the injury itself, but rather the impaired kidney function resulting from the injury. Thus, creatinine serves as a marker of kidney function rather than kidney injury, with elevated levels often appearing one or more days after the injury occurs. Additionally, creatinine levels are influenced by other factors unrelated to kidney function, such as an individual's muscle mass.

Urine output changes earlier than creatinine levels in cases of kidney injury and is easy to measure in intensive care patients, most of whom have urinary catheters. Reduced urine output is associated with an increased risk of mortality in intensive care patients, even when creatinine levels are normal. KDIGO defines reduced urine output as less than 0.5 milliliters of urine per kilogram of body weight per hour. However, this definition, which is essentially based on older studies of normal physiology, has been questioned in recent years. Reduced urine output is a normal physiological response to stress, such as surgery, making it challenging to distinguish physiological reductions in urine output from AKI. Several modern studies in surgical and intensive care contexts suggest that urine output lower than 0.5 ml/kg/h does not increase the risk of AKI or mortality. Based on these findings, lower thresholds have been proposed as a definition of AKI. More knowledge and studies that consider factors beyond urine output are needed to validate these findings. For instance, we lack knowledge about whether the relationship between urine output and patient outcomes is influenced by diuretic therapy, the amount of fluid administered, or fluid balance.

This research project aims to identify a possible threshold for urine output that reliably indicates AKI. The goal is also to examine the relationship between urine output and the severity of AKI, the need for renal replacement therapy (dialysis), long-term effects on kidney function, and mortality risk.

All adult patients treated in the intensive care unit at Uppsala University Hospital between 2016 and 2024 (up to the start of the study) will be included. Patients are identified through the Patient Administrative System for Intensive Care Units (PasIva). PasIva is an administrative support system used to report data to the Swedish Intensive Care Registry (SIR). Local data may need to be supplemented with information from SIR if necessary. The system provides data on reasons for ICU admission, severity of illness upon admission, interventions during intensive care, and 30- and 90-day mortality. Data in PasIva cannot be uploaded unless it is registered and formatted according to SIR's templates, ensuring validity.

From the local system Metavision, an electronic medical record system used in anesthesia and intensive care (Patient Data Management System, PDMS), data is retrieved on physiological variables such as urine output, fluid balance, body weight, medication, and organ-supportive treatments like renal replacement therapy (dialysis). Data is entered into Metavision hourly by ICU staff, ensuring high-resolution records. All medications administered in the relevant units are prescribed in Metavision.

From the medical record system COSMIC and databases managed by the Academic Laboratory at Uppsala University Hospital, data is collected on previous medical conditions, blood test results such as creatinine, and findings from diagnostic examinations. The Academic Laboratory is quality assured and accredited by SWEDAC according to SS-EN ISO 15189.

Patient data from the above sources will be merged to enable analysis. Data will be reviewed using standard procedures (e.g., measures of dispersion, plots) to detect anomalies indicative of errors in registration. We plan to divide the cohort into a subset for analysis and another for validation of the results. Multivariable statistical models will be applied to address the scientific questions described above.

ELIGIBILITY:
Inclusion Criteria:

* Admittance to intensive care units at Uppsala University Hospital between 2016-2024

Exclusion Criteria:

* Minimum age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients (>17 years of age) who have received care in the intensive care unit at Akademiska Sjukhuset since the implementation of the Metavision (an electronic medical record system used in anesthesia and intensive care (Patient Data Management System, PDMS)) from 2016-2017 (depending on the unit) up until the study start in 2024. To enable subgroup analyses and improve the reliability of estimates, the largest possible cohort is desired.
  Children will not be included in the study, as their urine production and normal reference values for blood markers of kidney function vary with age and differ from those of adults.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury according to KDIGO creatinine criteria. | Seven days rolling window.
  AKI by creatinine criteria is defined as any of the following: 1) Increase in SCr by ≥26.5 umol/l within 48 hours; or 2) Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days.
  Further, the severity of AKI is staged in 3 levels: 1) SCr 1.5-1.9 times baseline OR ≥26.5 umol/l increase; 2) SCr 2.0-2.9 times baseline; 3) SCr 3.0 times baseline OR increase in serum creatinine to ≥353.6 umol/l OR initiation of renal replacement therapy

IPD SHARING:
Plan to Share IPD: No
We are not allowed to share individual patient data according to decision in Swedish Ethical Review Authority. If a third party upon reasonable request present a valid authorization from the responsible government agency we might be allowed to share the data if we submit an amendment to the Swedish Ethical Review Authority.